CLINICAL TRIAL: NCT01373892
Title: Prospective, Randomised Study: Metabolic and Functional Effects of Bariatric Surgery Accessed Using PET and MRI
Acronym: Sleevepet2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Pirjo Nuutila, professor, cheif physician, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Sleevepet2
Record Dates: First submitted 2011-06-07; First posted 2011-06-15 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Masking Description: Sleeve or gastric bypass operation for obese
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Active Comparator): Slevve vs. Roux-Y
  Interventions: Procedure: Bariatric surgery
- Healthy lean volunteers (No Intervention)

INTERVENTIONS:
Procedure: Bariatric surgery
  Arms: Surgery

SUMMARY:
The objectives of this study are to measure effect of obesity on brain structure and molecular pathways, food-stimuli mediated brain activation response, on hormones affecting both feeding and energy balance as well as on bone metabolism and bone marrow fat. In the first phase the studies are performed at baseline before bariatric surgery and in the second phase post-operatively after 6 months. Regional free fatty acid uptake are studied with PET and 14(R, S)-[18F]-fluoro-6-thia-heptadecanoic acid ([18F]FTHA). Changes in body fat distribution are investigated with magnetic resonance imaging (MRI) Brain reward system response to food stimuli is assessed using functional MRI (fMRI) and white and grey matter volumes using diffusion tensor imaging (DTI). Brain neurotransmitter system will be measured with [11C]raclopride and [11C]carfentanil and PET. In the second part of the study the same variables are studied after bariatric surgery: either laparoscopic sleeve gastrectomy or Roux-en-Y gastric bypass.

DETAILED DESCRIPTION:
Regional free fatty acid uptake in myocardium, skeletal muscle, subcutaneous fat, visceral fat, pancreas, liver, brain, intestine and the bone are studied with PET and 14(R, S)-[18F]-fluoro-6-thia-heptadecanoic acid ([18F]FTHA). Changes in body fat distribution are investigated with magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS). Brain reward system response to food stimuli is assessed using functional MRI (fMRI) and white and grey matter volumes using diffusion tensor imaging (DTI).

The study consists totally of 60 study subjects. Of these 40 are morbidly obese adults, BMI

ELIGIBILITY:
Inclusion Criteria:

* 1) BMI > 40 kg/m2 or

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Tissue metabolism among morbidly obese persons assessed using PET, MRI and fMRI | Imaging studies will be performed before the bariatric surgery (day 1) and 6 months after. Healthy volunteers will be studied only once.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku PET Centre, Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dadson P, Honka MJ, Suomi T, Rokka A, Kauhanen S, Salminen P, Helmio M, James P, Elo LL, Olkkonen VM, Nuutila P. Characterization of Visceral Adipose Tissue Proteome Reveals Metabolic Changes and Inflammatory Signatures in Severe Obesity. Obesity (Silver Spring). 2026 Jan;34(1):127-137. doi: 10.1002/oby.70041. Epub 2025 Oct 12. PMID 41077621
- [Derived] Dadson P, Rebelos E, Jaakkola MK, Monfort-Pires M, Ojala R, Honka H, Kalliokoski KK, Klen R, Nuutila P, Ivaska KK. Differential associations of subcutaneous and visceral fat with bone turnover markers: A study on bariatric surgery patients with severe obesity and individuals without obesity. Int J Obes (Lond). 2025 Dec;49(12):2494-2502. doi: 10.1038/s41366-025-01888-1. Epub 2025 Aug 26. PMID 40854969
- [Derived] Dadson P, Honka MJ, Suomi T, Haridas PAN, Rokka A, Palani S, Goltseva E, Wang N, Roivainen A, Salminen P, James P, Olkkonen VM, Elo LL, Nuutila P. Proteomic profiling reveals alterations in metabolic and cellular pathways in severe obesity and following metabolic bariatric surgery. Am J Physiol Endocrinol Metab. 2025 Mar 1;328(3):E311-E324. doi: 10.1152/ajpendo.00220.2024. Epub 2025 Jan 17. PMID 39819027
- [Derived] Dadson P, Rebelos E, Honka H, Juarez-Orozco LE, Kalliokoski KK, Iozzo P, Teuho J, Salminen P, Pihlajamaki J, Hannukainen JC, Nuutila P. Change in abdominal, but not femoral subcutaneous fat CT-radiodensity is associated with improved metabolic profile after bariatric surgery. Nutr Metab Cardiovasc Dis. 2020 Nov 27;30(12):2363-2371. doi: 10.1016/j.numecd.2020.07.010. Epub 2020 Jul 15. PMID 32919861
- [Derived] Savolainen AM, Karmi A, Immonen H, Soinio M, Saunavaara V, Pham T, Salminen P, Helmio M, Ovaska J, Loyttyniemi E, Heiskanen MA, Lehtimaki T, Mari A, Nuutila P, Hannukainen JC. Physical Activity Associates with Muscle Insulin Sensitivity Postbariatric Surgery. Med Sci Sports Exerc. 2019 Feb;51(2):278-287. doi: 10.1249/MSS.0000000000001778. PMID 30247434
- [Derived] Immonen H, Hannukainen JC, Kudomi N, Pihlajamaki J, Saunavaara V, Laine J, Salminen P, Lehtimaki T, Pham T, Iozzo P, Nuutila P. Increased Liver Fatty Acid Uptake Is Partly Reversed and Liver Fat Content Normalized After Bariatric Surgery. Diabetes Care. 2018 Feb;41(2):368-371. doi: 10.2337/dc17-0738. Epub 2017 Nov 20. PMID 29158250
- [Derived] Honka H, Koffert J, Hannukainen JC, Tuulari JJ, Karlsson HK, Immonen H, Oikonen V, Tolvanen T, Soinio M, Salminen P, Kudomi N, Mari A, Iozzo P, Nuutila P. The effects of bariatric surgery on pancreatic lipid metabolism and blood flow. J Clin Endocrinol Metab. 2015 May;100(5):2015-23. doi: 10.1210/jc.2014-4236. Epub 2015 Mar 3. PMID 25734253
- [Derived] Tuulari JJ, Karlsson HK, Hirvonen J, Salminen P, Nuutila P, Nummenmaa L. Neural circuits for cognitive appetite control in healthy and obese individuals: an fMRI study. PLoS One. 2015 Feb 6;10(2):e0116640. doi: 10.1371/journal.pone.0116640. eCollection 2015. PMID 25658479
- [Derived] Honka H, Hannukainen JC, Tarkia M, Karlsson H, Saunavaara V, Salminen P, Soinio M, Mikkola K, Kudomi N, Oikonen V, Haaparanta-Solin M, Roivainen A, Parkkola R, Iozzo P, Nuutila P. Pancreatic metabolism, blood flow, and beta-cell function in obese humans. J Clin Endocrinol Metab. 2014 Jun;99(6):E981-90. doi: 10.1210/jc.2013-4369. Epub 2014 Feb 14. PMID 24527718